CLINICAL TRIAL: NCT05746130
Title: A Comparison of the Effects of a Plastic-Free Nutrition Program, Interactive Education, and Exposure Feedback on Bisphenol-A Levels in Adolescents With Packaged Product High Usage
Brief Title: Effect of Preventive Education on Reducing Urinary Bisphenol-A Levels in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma Ulusoy, PhD student, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TDK-2023-6207
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Behavior; Bisphenol A; Urine
Keywords: Bisphenol A; urinary test; adolescent; Packaged Product Usage
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Nonrandomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- plastic-free diet program (Experimental): Plastic-free nutrition program will include plastic-free diet, peer mentoring, interactive education and BPA exposure feedback.
  Interventions: Behavioral: Plastic-free diet program; Behavioral: Plastic-free diet education program; Behavioral: BPA exposure feedback
- plastic free diet education program (Active Comparator): This group will take peer mentoring, interactive education and BPA exposure feedback.
  Interventions: Behavioral: Plastic-free diet education program; Behavioral: BPA exposure feedback
- BPA exposure feedback (Active Comparator): This group will take only BPA exposure feedback.
  Interventions: Behavioral: BPA exposure feedback

INTERVENTIONS:
Behavioral: Plastic-free diet program — Applying the plastic-free diet as four meals (three main meals, one snack) in pension kitchen. Promoting of glass water bottle giving and daily use.
  Interactive education program: Slogan competition, school board preparation, short film shooting, school canteen visits and plastic-free nutrition day event with the adolescents for four weeks by the researcher.
  Peer education will doing by Adolescents with Packaged Product Low Usage Feedback about BPA levels in theirs urinary sample.
  Arms: plastic-free diet program
Behavioral: Plastic-free diet education program — Interactive education program: Slogan competition, school board preparation, short film shooting, school canteen visits and plastic-free nutrition day event with the adolescents for four weeks by the researcher.
  Peer education will doing by Adolescents with Packaged Product Low Usage Feedback about BPA levels in theirs urinary sample
  Arms: plastic free diet education program; plastic-free diet program
Behavioral: BPA exposure feedback — Feedback about BPA levels in theirs urinary sample

SUMMARY:
It is known that Bisphenol-A (BPA) is the endocrine disrupting chemical that is most exposed by oral intake in daily life. Critical life periods when the sensitivity to these substances is known to be maximum; prenatal, postnatal and adolescence periods. The aim of this study is to compare the effects of plastic-free nutrition program, interactive education and BPA exposure feedback on urinary Bisphenol-A levels in adolescents with high use of packaged products.

DETAILED DESCRIPTION:
By simple random sampling, female adolescents (n=36) staying in a high school hostel will be the intervention group, female adolescents not staying in hostels (n=36) will be the first comparison group, and female adolescents from another high school (n=36) will be the second comparison group. Plastic-free nutrition program (plastic-free diet, peer mentoring, interactive education and BPA exposure feedback) will be applied to the intervention group. Interactive training and BPA exposure feedback will be given to comparison group one, while only BPA exposure feedback will be given to comparison group two. Before and after the interventions, urinary BPA levels, use of plastic packaged products and bad nutrition attitudes of the adolescents will be monitored.

ELIGIBILITY:
Inclusion Criteria:

Willingness to participate in the research Being in the 14-18 age group Being a female student High (61-80 points) or moderate-high (41-60 points) scores from the plastic packaged product use questionnaire (PAUKA) Having a smart mobile phone Absence of obesity, hypertension, diabetes mellitus, cardiovascular, asthma, thyroid and kidney dysfunction or disease Absence of any syndrome (Metabolic, Turner Rett and Down syndrome etc.) Absence of any medication used continuously Absence of any chronic disease reported by the physician in the student follow-up/examination report

Exclusion Criteria:

Leaving school and hostel Not giving a spot urine sample Not participating in the plastic-free diet program in the hostel for the last week.

Desire to leave the study Participation in trainings <50% Diagnosis of disease (diabetes mellitus, kidney disease, gluten or lactose intolerance, etc.) in which dietary habits were changed during the study.

Experiencing a mental or physical illness that will prevent the continuity of participation in the study.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Urinary BPA level | Baseline-Second month
  Urinary Bisphenol A

SECONDARY OUTCOMES:
Plastic Packaged Product Usage | Baseline-Second month
  0-20 points indicate the use of low plastic packaged products, 21-40 points indicate the use of medium plastic packaged products, 41-60 points indicate the use of medium-high plastic packaged products, and 61-80 points indicate the use of high plastic packaged products.
Attitude Towards Healthy Eating | Baseline-Second month
  11 points obtained from the scale are very low, 12-22 points low, 23-33 points medium, 34-44 points high, 45-55 points ideally high, indicating the attitude towards healthy and plastic-free nutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Döşemealtı Mesleki ve Teknik Anadolu Lisesi, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided